CLINICAL TRIAL: NCT02856048
Title: Assessment of the Effect of a Co-treatment With GnRH Analogs on the Ovarian Reserve in Adolescents and Young Women Treated With Alkylating Agents for Cancer
Brief Title: Co-treatment With GnRH Analogs on the Ovarian Reserve in Young Women Treated With Alkylating Agents for Cancer
Acronym: PRESOV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140932; 2015-001121-17 (EudraCT Number)
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Cancer; Toxicity Due to Chemotherapy; Sarcoma; Osteosarcoma; Lymphoma; Ewing Sarcoma
Keywords: GnRH agonist; Ovarian reserve; Fertility Preservation; Alkylating Agents
MeSH Terms: conditions — Neoplasms; Sarcoma; Osteosarcoma; Lymphoma; Sarcoma, Ewing | interventions — Triptorelin Pamoate; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptorelin (GnRHa) + Chemotherapy (Experimental): Triptorelin LP 3 mg (DECAPEPTYL LP 3 mg, IPSEN) 3 mg every 28±3 days, intramuscular during chemotherapy
  Interventions: Drug: Triptorelin (GnRHa) + Chemotherapy
- Chemotherapy alone (No Intervention): Patient having a chemotherapy without drug injection for fertility preservation

INTERVENTIONS:
Drug: Triptorelin (GnRHa) + Chemotherapy — During her chemotherapy, the patient in the experimental arm will have regular injections of Triptorelin (DECAPEPTYL LP 3 mg, IPSEN) in order to preserve her fertility
  Other Names: GnRH Agonist injections
  Arms: Triptorelin (GnRHa) + Chemotherapy

SUMMARY:
The purpose of this study is to determine the efficacy of a temporary ovarian suppression obtained by administration of a gonadotropin releasing hormone agonist during alkylating agents containing chemotherapy on ovarian reserve assessed by Anti-Müllerian hormone (AMH) serum levels in adolescents and young women with cancer.

DETAILED DESCRIPTION:
This is a French, Prospective, Multicentre, Open, Randomised study To determine the efficacy of a temporary ovarian suppression obtained by administration of a Gonadotropin Releasing Hormone agonist (GnRHa) on maintaining ovarian reserve, patients will be randomized, half of them receiving Triptorelin extended release (LP) 3 mg intramuscularly every 28±3 days, starting at the inclusion visit and at least 72 days before chemotherapy with alkylating agents until 1 month after end of chemotherapy (mean duration: 12 months).

The primary objective of the study is to determine the effect of a temporary ovarian suppression achieved through administration of a gonadotropin releasing hormone agonist (triptorelin LP 3 mg) during alkylating agents containing chemotherapy on ovarian reserve assessed by AMH serum levels in adolescents and young women with cancer.

Number of centres 19 Research period

* Recruitment duration 2 years
* The duration of participation of each patient is: 3 years
* The duration of the treatment period is: 1 year
* The duration of the follow-up period is: 2 years
* Total duration: 5 years

Statistical analysis:

1. Sample size and design One Hundred and sixty (160) patients will be included in this study in order to ensure at least 128 patients who will complete the study.

   This number of patients should allow us to identify with a power of 80 % a difference of 5 pmol/L in AMH serum levels between the two groups, when accepting a risk alpha of 0.05.
2. Analysis populations The main analysis will be an intention-to-treat (ITT) analysis, which will be performed on all the randomized patients with a value of the main criterion of judgment (AMH level at M24). A per-protocol (PP) analysis will also be performed, as a secondary analysis, excluding patients with major protocol deviation defined a priori.
3. Primary criteria The value of AMH level at month 24will be compared between the two treatment groups using a test t of Student if AMH values are normally distributed and a non-parametric Wilcoxon test if not.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 12 to 25 years
* Puberty Tanner 2 or more
* Diagnosis of cancer: Sarcoma, Ewing, Osteosarcoma, Lymphoma
* Chemotherapy protocol with alkylating agents at an intermediate ovarian toxicity risk (Cyclophosphamide 6 g/m2, Ifosfamide 50 g/m2, Procarbazine 4 g/m2, Lomustine 350 mg/m2 or Melphalan 140 mg/m2 or a combination of these drugs).
* All patients with an osteosarcoma, Ewing sarcoma excepted pelvic localisation, Hodgkin lymphoma treatment group III (stages II B, III B and IV), B cell lymphoma group C, rhabdomyosarcoma treated with at least 8 Ifosfamide Vincristin Actinomycin (IVA) courses, synoviosarcoma group II T>5 cm and group III, adult type sarcoma group I and II T>5 cm and group III.
* Before starting any chemotherapy
* Covered by a medical insurance

Exclusion Criteria:

* Prepubertal
* Pregnant
* Planned brain or pelvic radiotherapy
* Planned stem cell transplantation
* Ovariectomy
* Having already received chemotherapy with alkylating agents
* Hypersensitivity to any component of GnRHa

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Variation in AMH serum levels between both groups | at 24 months
  Centralised hormonal dosages

SECONDARY OUTCOMES:
Number of patients with AMH serum levels < 5th percentile in each group | at 24 months
Intra-patient variation in AMH serum levels between groups | up to 36 months
  Centralised hormonal dosages and study of potential factors associated with the efficacy of GnRHa co-treatment in preventing ovarian reserve loss (if there is one)
Antral Follicular Count (AFC) on ultrasound between the 2 groups | at month 24
  centralised blind evaluation by an independent reader on compact disc (CD) registration of AFC
Delay of resumption of menses between the 2 groups | up to the end of the follow up (an average of 3 years)
  Comparison of delay of resumption of menses between the 2 groups
Levels of markers of ovarian reserve: AMH, Follicle-stimulating hormone (FSH), Estradiol between groups | at months 12, 24 and 36
  Centralised hormon dosage
Pregnancy rate in the 2 groups | up to the end of the follow up (an average of 3 years)
Adverse events related to Triptorelin co-treatment | up to the end of the follow up (an average of 3 years)
Relative change in Bone Mass Density (BMD) of the lumbar spine, left femoral neck and whole body in the 2 groups | at the baseline and at month 12 and month 36
  centralised blind evaluation by an independent reader on CD registration of BMD assessed by dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Cecile THOMAS-TEINTURIER, MD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No